CLINICAL TRIAL: NCT05149014
Title: Real-world Study on Safety, Effectiveness and Quality of Life of Trastuzumab Deruxtecan in Patients with Metastatic or Unresectable HER2-positive Breast Cancer: a French Ambispective Multicentre 2 Year-follow-up Cohort Study
Brief Title: Safety, Effectiveness and Quality of Life of Trastuzumab Deruxtecan in Patients with HER2+ Breast Cancer
Status: Completed | Type: Observational
Sponsor: Daiichi Sankyo France (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-A02007-34
Record Dates: First submitted 2021-11-25; First posted 2021-12-08 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: HER2-positive Breast Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Collection of data in real life conditions on satefy, effectiveness and quality of life of trastuzumab deruxtecan in patients with metastatic or unresectable HER2-positive breast cancer.

DETAILED DESCRIPTION:
The present observational study aims to collect data on long-term safety of trastuzumab deruxtecan, with a primary endpoint on trastuzumab deruxtecan related adverse drug reactions (ADRs) of interest. Data on patient profile, treatment history (before, during and after trastuzumab deruxtecan administration), effectiveness and health-related quality of life will also be collected in a real-life setting, to confirm and complement data from clinical trials. Patients will be recruited whether they have started trastuzumab deruxtecan treatment or will start it at the time of inclusion, whether they were prescribed compassionate trastuzumab deruxtecan or marketed Enhertu®, in order to rapidly collect a large set of data.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult patient (age ≥ 18 years);
* Unresectable or metastatic HER2+ breast cancer, previously treated with at least 2 lines of anti-HER2, and:

  * previously treated by compassionate trastuzumab deruxtecan (ATU group), or
  * previously treated or planned to be treated by trastuzumab deruxtecan (Enhertu®), upon the investigator's decision (Post-Marketing authorization group);
* Patient who expresses non-opposition to participate in the study, or deceased patient who did not express his/her opposition to the use of his/her personal data while alive.

Exclusion Criteria:

- Previous participation in an interventional clinical trial with trastuzumab deruxtecan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Unresectable or metastatic HER2+ breast cancer, treated at least once with trastuzumab deruxtecan
Sampling Method: Probability Sample
Enrollment: 306 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with at least one Trastuzumab deruxtecan related Adverse Drug Reaction of interest | 2 years following the start of administration of Trastuzumab deruxtecan
  The primary endpoint is the percentage of patients with at least one Trastuzumab deruxtecan related Adverse Drug Reaction of interest

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique des Flandres, Coudekerque-Branche, France